CLINICAL TRIAL: NCT07144709
Title: A 6-months Prospective, Observational Study to Evaluate the Quality of Life of Patients Treated With Phytotherapy or Alpha-blockersfor Benign Prostatic Hyperplasia
Brief Title: A 6-months Observational Study to Evaluate the Quality of Life of Patients Treated With Phytotherapy or Alpha-blockers for Benign Prostatic Hyperplasia
Acronym: PERQoL
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Kappa Santé (Industry)
Responsible Party: Sponsor
Other Study IDs: PierreFabreMed
Record Dates: First submitted 2025-07-23; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Phytotherapy; Adrenergic alpha-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phytotherapy: Patients initiating a first-line phytotherapy treatment for LUTS/BPH in monotherapy
  Interventions: Drug: Phytotherapy
- Alpha-blockers: Patients initiating a first-line alpha-blockers treatment for LUTS/BPH in monotherapy

INTERVENTIONS:
Drug: Phytotherapy — Phytotherapy or alphablockers
  Other Names: Alpha-blockers
  Groups: Phytotherapy

SUMMARY:
This is a prospective, multicentre, non-interventional study, conducted in France and Spain, in primary care practices and designed to assess the QoL of patients under phytotherapy or alpha-blockers for LUTS/BPH. The study will not provide or recommend any treatment or procedure.

DETAILED DESCRIPTION:
Any patient with moderate to severe LUTS/BPH initiating treatment with PT or AB during the inclusion period will be invited to participate in the study. Per usual practice, the physician will prescribe a treatment independently of the study. Patients will be consecutively enrolled in each of the 2 groups (PT or AB), regardless of the number of patients already enrolled in the other group. An average of 6 patients per General Practitioner (GP) is expected, i.e. 3 patients in each group. A GP who has reached 3 patients in a group will continue to recruit in the second group until reaching 2 groups of 3 patients. Once the two groups of 3 patients have been completed, the inclusions may be re-opened following the same procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Age ≥ 40 years at the time of enrolment
* Diagnosed with moderate to severe LUTS/BPH (IPSS ≥ 12)
* Initiating a first-line PT or AB treatment for LUTS/BPH in monotherapy
* Provided informed consent or non-opposition to study inclusion, and for the use of data, according to local regulations

Exclusion Criteria:

* Underwent prostate surgery or urinary tract surgery
* Diagnosed with one or several other diseases involving urinary function or prostate Diagnosed with BPH with complications (recurrent urinary tract infection, recurrent acute urinary retention, bladder calculus, bladder diverticulum, hydronephrosis, overflow incontinence, recurrent hematuria, obstructive renal failure) Participating in interventional trial on any investigational drug at time of inclusion Under treatment of the urinary functions

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating sites will be encouraged to propose the study to all patients meeting the eligibility criteria, in a consecutive manner, when they come for consultation, in order to minimize bias in patient selection.Each investigator site will include the samenumber of patients initiating PT and initiating AB.Treatment choice should be made by the investigator as routine practice. No medical therapy is required for this study.Investigators should ensure that IPSS total score meets the eligibility criteria before enrolling patients in the study.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Benign Prostatic Hypertrophy Health-Related Quality of Life Questionnaire (BPHQOL9) M6 | 6 months
  Mean difference in BPHQOL9 scores between baseline and M6, by group of treatment (PT and AB).
  For BPHQOL9, the total score can range from 0 to 90 (sum of all 9 items). A higher score means a better quality of life.

SECONDARY OUTCOMES:
Benign Prostatic Hypertrophy Health-Related Quality of Life Questionnaire (BPHQOL9), M6 | 6 months
  Mean difference in BPHQOL9 scores between baseline and M3 or M6, by group of treatment For BPHQOL9, the total score can range from 0 to 90 (sum of all 9 items). A higher score means a better quality of life.
Quality of life Benign Prostatic Hypertrophy Health-Related Quality of Life Questionnaire (BPHQOL9) | 6 months
  Quality of life changes using BPHQOL9 questionnaire over the 6-month period.
  For BPHQOL9, the total score can range from 0 to 90 (sum of all 9 items). A higher score means a better quality of life.
Urinary symptoms profiles | 6 months
  Urinary symptoms profiles using International Prostate Score Symptom (IPSS) questionnaire over the 6-month period by group of treatment.
  Score has a total range from 0 to 35 (sum of the first 7 questions) with 3 defined severity states (0-7 = mild; 8-19 = moderate; 20-35 = severe). A higher score means a worse urinary difficulties.
Sexual Fonction | 6 months
  Sexual function and satisfaction using Male Sexual Health Questionnaire (MSHQ) over the 6-month period by group of treatment.
  The MSHQ total score ranges from 0 to 125 (sum of all items). Higher scores indicate better sexual function.
Safety (Adverse events) | 6 months
  Safety assessment over the 6-month period by group of treatment

OTHER OUTCOMES:
Correlation | 6 months
  BPHQOL9 total score and IPSS QoL score will be estimated per patient at each time measurement (baseline, M3 and M6) in order to assess corelations between both scores

CONTACTS AND LOCATIONS:
Overall Officials: EID, Study Director — Pierre Fabre Laboratories
Locations (31):
- France (20):
  - Medical Office of Delsart MD, Bersée
  - Medical Office of Breton MD, Béziers
  - Medical Office of Guiu MD, Ferrals-les-Corbières
  - Medical Office of Patron MD, Gap
  - Medical Office of Coulon MD, Giromagny
  - Medical Office of Dassa MD, Istres
  - Medical Office of Rigaud MD, Lamagistère
  - Medical Office of Specht MD, Lambersart
  - Medical Office of Mesguich MD, Le Blanc-Mesnil
  - Medical Office of Dassonval MD, Marles-les-Mines
  - Medical Office of Cayron MD, Montpellier
  - Medical Office of Chassagne MD, Montpellier
  - Medical Office of Baranes MD, Paris
  - Medical Office of Labregere MD, Paris
  - Medical Office of Merlin MD, Raimbeaucourt
  - Medical Office of Lemercier MD, Royan
  - Medical Office of Margueritte MD, Six-Fours-les-Plages
  - Maison de Santé MEDIVIE, Templeuve-en-Pévèle
  - Medical Office of Demoulin MD, Val-de-Vesle
  - Medical Office of David MD, Verzy
- Spain (11):
  - Cs Vargas, Santander, Santander, Cantabria
  - C.S. San Jose, A Coruña
  - C.S. Zona Ii, Albacete
  - C.S. Aldea Moret, Cáceres
  - C.S. Fuencarral, Madrid
  - C.S. Mendiguchia, Madrid
  - Centro Urología, Andrología Y Salud Sexual, Palma de Mallorca
  - C.S. Rotxapea, Pamplona
  - C.S. Soria Rural, Soria
  - C.S. Laguna de Duero, Valladolid
  - Cs Villamayor de Gallego, Zaragoza

IPD SHARING:
Plan to Share IPD: No